CLINICAL TRIAL: NCT01179529
Title: Single- Arm Trial to Identify Potential Markers Underlying Variability in Response to Omalizumab (Xolair®) Treatment in Atopic Dermatitis
Brief Title: Atopic Dermatitis Biomarker Identification Trial in Omalizumab Usage
Acronym: AMB-WEI-1052-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: AMBITIOUS
Record Dates: First submitted 2010-08-02; First posted 2010-08-11 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Atopic Dermatitis; Atopic Eczema
Keywords: Atopic dermatitis (atopic eczema)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omalizumab (Experimental)
  Interventions: Drug: Omalizumab (Xolair®)

INTERVENTIONS:
Drug: Omalizumab (Xolair®)

SUMMARY:
This study aims at evaluating the therapeutic potential of omalizumab in atopic dermatitis, and to work out biomarkers predictive of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18-70 years of age, body weight ≥ 20 kg and ≤ 150 kg
* Dermatological diagnosis of AD, SCORAD >=20
* A positive RAST (≥CAP1) result for at least one aeroallergen specific IgE and total IgE >=100kU/l at screening (or within the previous 12 months)
* Eligible to receive systemic therapy for AD in accordance to local guidelines
* Signed informed consent from patient

Exclusion Criteria:

* Evidence of skin disease other than AD (e.g. psoriasis) at the inclusion time
* Treatment with systemic AD medications or any investigational drug within a 30-day washout period
* Concomitant treatment with substances interfering with the immune system
* Permanent severe diseases, especially those affecting the immune system, except asthma
* Pregnancy or breast feeding
* History of food or drug related severe anaphylactoid or anaphylactic reaction(s)
* History or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia
* History or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy
* Elevated serum IgE levels for reasons other than allergy and/or urticaria (e.g.: parasite infections, hyperimmunoglobulin E syndrome, Wiskott - Aldrich syndrome or clinical allergic bronchopulmonary aspergillosis)
* Evidence of severe renal dysfunction or significant hepatic disease
* Evidence for active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
* History of malignancy of any organ system, treated or untreated, whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin
* Clinically significant laboratory abnormalities (not associated with AD) at Visit 1
* Known hypersensitivity to any ingredients, including excipients (sucrose, histidine, polysorbate 20) of the study medication or drugs related to Omalizumab (e.g.: monoclonal antibodies, polyclonal gammaglobulin)
* Patients who are considered potentially unreliable or where it is envisaged the patient may not consistently attend scheduled study visits
* Patients with serious psychiatric and/or psychological disturbances
* Patients with a history of drug or alcohol abuse
* Patients who are unable to complete a patient diary or complete questionnaires on paper
* Patients with any other condition or prior/current treatment, which in the opinion of the investigator renders the patient ineligible for the study schedule

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
To evaluate efficacy of Omalizumab treatment in a sample of adult patients with moderate to severe AD

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Weidinger, Prof.Dr.med., Principal Investigator
Locations (1):
- Klinikum rechts der Isar Dermatologie/Biederstein, Munich, Bavaria, Germany